CLINICAL TRIAL: NCT06067971
Title: Evaluation of the Feasibility of Using Augmented Reality in Laparoscopic Surgery, by a Clinical Study During Gynecological Laparoscopic Surgical Procedures.
Acronym: ENDORA2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: RBHP 2021 CHAUVET; 2021-A01987-34 (Other: ANSM)
Record Dates: First submitted 2023-09-28; First posted 2023-10-05 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Myoma;Uterus; Adenomyoma of Uterus
Keywords: Augmented Reality; Laparoscopic surgery; Uterine myomectomy; Uterine adenomyomectomy; Hysterectomy; Minimally invasive surgery
MeSH Terms: conditions — Myofibroma | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Laparoscopic surgery with the augmented reality device (Experimental)
  Interventions: Device: Laparoscopic surgery with augmented reality device

INTERVENTIONS:
Device: Laparoscopic surgery with augmented reality device — Gynecological laparoscopic surgery with augmented reality device.

SUMMARY:
Augmented Reality is a technology that allows surgeons to superimpose virtual images from preoperative imaging onto the endoscopic vision system intraoperatively. The goal of this clinical trial is to demonstrate that the use of augmented reality during laparoscopic gynecological surgery with a dedicated device could provide assistance to the surgeon, in terms of technical comfort and better visualization of the benign tumor to be resected on a mobile organ.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 (included) and 84 (included),
* Patient with intrauterine myoma, with indication for surgical management by laparoscopic myomectomy, or uterine pathology with indication for surgical management by laparoscopic hysterectomy,
* Patient affiliated or beneficiary of a health insurance scheme,
* Patient agreeing to participate in the study after having received the written information document and signed the consent form.

Exclusion Criteria:

* Patients under 18 or over 84 years of age,
* Patients with contraindications to MRI (pacemaker, ocular metal splinters, etc.),
* Impossibility of planned surgery,
* Patient with endometrial cancer contraindicating laparoscopic surgery,
* Known pregnant or breast-feeding patient,
* Patient of legal age, under guardianship or curatorship,
* Patients whose regular follow-up is impossible for geographical, psychological, family or social reasons (these reasons will be collected).

Ages: 18 Years to 84 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-03-29 (Actual); Primary Completion 2025-04-16 (Actual); Study Completion 2025-05-15 (Actual)

PRIMARY OUTCOMES:
The feasibility of augmented reality will be measure using the SURG-TLX scale | In the intra-operative phase of the study
  The feasibility of the technique will be considered satisfactory if the SURG-TLX score given by the surgeon at the end of the procedure is less than or equal to 33.7 (threshold defined by experts).

SECONDARY OUTCOMES:
Score of the surgeon's performance in using the augmented reality device | In the intra-operative phase of the study
  Measuring the performance-related score when using the augmented reality device by filling in a scale.
Collection of operative time | In the intra-operative phase of the study
  Collection of operating times for the entire surgery, as well as the various times associated with augmented reality device installation.
Number of device failures during surgery | In the intra-operative phase of the study
  Number of device failures during surgery (defined as an abrupt stop of the device during its use)
Number of failures to start up the software | In the intra-operative phase of the study
  Collection of the number of failures to set up the augmented reality device
Collection of the real direct medical costs of the procedure from an institutional point of view. | From the date of the surgery to the date of the first post-operative visit, usually 1 month after the surgery
  Collection of the real direct medical costs of the procedure from an institutional point of view.
Number of laparoscopic/laparotomy conversions | In the intra-operative phase of the study
  Collection of the number of laparoscopic/laparotomy conversions.
Number of intraoperative and postoperative complications | From the date of the surgery to the date of the first post-operative visit, usually 1 month after the surgery
  Collection of the number of intraoperative and postoperative complications (especially vascular or ureteral wounds).
Quantification of bleeding | In the intra-operative phase of the study
  Collection of bleeding volume during the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Pauline CHAUVET, Principal Investigator — pchauvet@chu-clermontferrand.fr
Locations (3):
- France (3):
  - Polyclinique Urbain V, Avignon
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU de Saint-Étienne, Saint-Etienne